CLINICAL TRIAL: NCT00326976
Title: A Multicenter, Double Blind, Randomized, Placebo Controlled Study to Measure the Effect of FX06 (a Fibrin Derived Peptide Bbeta15-42) on Ischemia Reperfusion Injury in Patients Undergoing Primary Percutaneous Coronary Intervention (PCI): The "F.I.R.E." Study
Brief Title: Efficacy of FX06 in the Prevention of Myocardial Reperfusion Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fibrex Medical Research & Development GmbH (Industry)
Responsible Party: Dr: Rainer Henning, Fibrex Medical Research & Development GmbH
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FX06AQ-II-01
Record Dates: First submitted 2006-05-16; First posted 2006-05-17 (Estimated); Last update posted 2007-12-04 (Estimated); Status verified 2007-12

CONDITIONS: Myocardial Ischemia; Coronary Disease; Myocardial Infarction
Keywords: Angioplasty, Transluminal, Percutaneous Coronary; Myocardial Revascularization
MeSH Terms: conditions — Myocardial Ischemia; Coronary Disease; Myocardial Infarction | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 400 mg injected in 2 divided boluses
  Interventions: Drug: FX06; Procedure: Percutaneous coronary intervention
- 2 (Placebo Comparator): Matching placebo
  Interventions: Drug: FX06; Procedure: Percutaneous coronary intervention

INTERVENTIONS:
Drug: FX06 — 400 mg as intravenous injection in two divided boluses
Procedure: Percutaneous coronary intervention

SUMMARY:
The purpose of the study is to evaluate whether FX06 is capable of limiting infarct size following balloon catheterization for acute myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have given informed consent
* Patients after primary percutaneous coronary intervention (PCI) for acute ST-elevation myocardial infarction (STEMI)
* Men or women with no child bearing potential
* Onset of symptoms to balloon time < 6 hours
* ST-elevation of at least 2 mm in at least 3 leads on 12-lead electrocardiogram (ECG)
* Primary PCI indicated per standard of care
* First myocardial infarction (MI)
* Single index lesion with complete occlusion [thrombolysis in myocardial infarction (TIMI) flow 0/I] of one target vessel.

Exclusion Criteria:

* History of MI (from patient history, or from ECG)
* Chest pain or other angina symptoms in the 24 hours before the first recognized symptoms of the acute myocardial infarction (AMI)
* Need for coronary artery bypass graft (CABG)
* Administration of any thrombolytic agent since onset of AMI symptoms
* Serious procedural complications (e.g., procedural unintended occlusion of coronary artery branch, cardiac tamponade, emergency bypass operation, LM dissection, etc.)
* Presence of cardiogenic shock: hemodynamically unstable and/or need for positive inotropic agents
* Contraindication to cardiovascular magnetic resonance (CMR): claustrophobia, pacemakers, defibrillators and other electronic devices, and metallic cerebral clips; frequent extrasystoles (> 12/Min) or atrial fibrillation (AF).
* Known renal dysfunction defined as serum creatinine > 250 µmol/l
* Previous CABG
* History of congestive heart failure (CHF)
* Body mass index (BMI) > 35
* Patients who cannot communicate reliably with the investigator
* Patients who are unlikely to cooperate with the requirements of the study
* Patients who are unwilling and/or unable to give informed consent
* Patients at increased risk of death from a pre-existing concurrent illness
* Patients participating in another clinical study
* Patients who have used any other investigational drugs within 1 month of first dosing
* Patients who have participated already in this study
* Patients who are employees at the investigational site; relatives or spouse of the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2006-08; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Infarct size as measured by cardiac MRI | 5-7 days post intervention

SECONDARY OUTCOMES:
Myocardial scar mass and left ventricular function | 4 months post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Dan Atar, MD, Principal Investigator — Aker University Hospital, Oslo, Norway
Locations (32):
- Austria (2):
  - Allgemeines Krankenhaus Wien, Vienna
  - Wilhelminen-Spital, Vienna
- Belgium (2):
  - Academisch Ziekenhuis van de vrije Universiteit, Brussels
  - Cliniques Universitaires St-Luc, Brussels
- Czechia (2):
  - I. Interna Klinika, Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Kardiologicke oddeleni, Masarykova nemocnice, Ústí nad Labem
- Amtssygehuset i Gentofte, Hellerup, Denmark
- Germany (15):
  - Universitätsklinikum Aachen, Aachen
  - Zentralkliniken Bad Berka, Bad Berka
  - Charite, Campus Benjamin Franklin, Berlin
  - Vivantes Klinikum Neukölln, Klinik für Innere Medizin, Berlin
  - Ev. Freikirchliches KH Bernau und Herzzentrum Brandenburg, Bernau
  - Krankenhaus Düren gem. GmbH, Innere I (Kardiologie), Düren
  - Universitätsklinikum Freiburg - Innere Medizin III, Freiburg im Breisgau
  - Krankenhaus Martha-Maria Halle-Dölau - Innere Medizin I, Halle
  - Martin-Luther-Universität Halle-Wittenberg, Klinikum der Medizinischen Fakultät, Inner Medizin III, Halle
  - Universitätsklinikum Schleswig-Holstein-Klinik f. Kardiologie, Kiel
  - Universität Leipzig, Klinik für Innere Medizin, Herzzentrum, Leipzig
  - Universitätsklinikum Schleswig-Holstein,Medizinische Klinik II, Campus Lübeck, Lübeck
  - Universitätsklinikum Mannheim, I. Medizinische Klinik, Mannheim
  - Deutsches Herzzentrum München, Munich
  - Klinik für Innere Medizin und Kardiologie, Marienhospital Osnabrück, Akademisches Lehrkrankenhaus der Medizinischen Hochschule Hannover, Osnabrück
- Vilnius University Hospital "Santariskiu klinikos", Center of Cardiology and Angiology, Vilnius, Lithuania
- Netherlands (2):
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - St. Antonius Ziekenhuis, Nieuwegein
- Poland (3):
  - Krakowski Szpital Specjalistyczny im. Jana Pawla II, Krakow
  - Zaklad Szybkiej Diagnostyki, Kardiologicznej, Szpital im. Biekalskiego, Lodz
  - Samodzielny Publiczy, Zaklad Opieki Zrowotnej, Uniwersytecki Szpital Kliniczny Nr. 3, Im. dr Seweryna Sterlinga, Lodz
- Institute for Cardiovascular Disease, Timișoara, Romania
- Sweden (2):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Universitetssjukhuset, Linköping
- Universitätshospital Zürich, Zurich, Switzerland

REFERENCES:
- [Derived] Hallen J, Jensen JK, Fagerland MW, Jaffe AS, Atar D. Cardiac troponin I for the prediction of functional recovery and left ventricular remodelling following primary percutaneous coronary intervention for ST-elevation myocardial infarction. Heart. 2010 Dec;96(23):1892-7. doi: 10.1136/hrt.2009.190819. PMID 21062778
- [Derived] Hallen J, Petzelbauer P, Schwitter J, Geudelin B, Buser P, Atar D. Impact of time to therapy and presence of collaterals on the efficacy of FX06 in acute ST elevation myocardial infarction: a substudy of the F.I.R.E., the Efficacy of FX06 in the prevention of myocardial reperfusion injury trial. EuroIntervention. 2010 Apr;5(8):946-52. PMID 20542780
- [Derived] Atar D, Petzelbauer P, Schwitter J, Huber K, Rensing B, Kasprzak JD, Butter C, Grip L, Hansen PR, Suselbeck T, Clemmensen PM, Marin-Galiano M, Geudelin B, Buser PT; F.I.R.E. Investigators. Effect of intravenous FX06 as an adjunct to primary percutaneous coronary intervention for acute ST-segment elevation myocardial infarction results of the F.I.R.E. (Efficacy of FX06 in the Prevention of Myocardial Reperfusion Injury) trial. J Am Coll Cardiol. 2009 Feb 24;53(8):720-9. doi: 10.1016/j.jacc.2008.12.017. PMID 19232907